CLINICAL TRIAL: NCT01143792
Title: Evaluation of Treatments for Homeless Youth: CRA, MET and Case Management
Brief Title: Evaluation of Treatments for Homeless Youths
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Natasha Slesnick, Ph.D., Ohio State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2005B0078; R01DA013549 (NIH)
Record Dates: First submitted 2010-06-11; First posted 2010-06-14 (Estimated); Results first posted 2013-04-16 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Substance Abuse
Keywords: Substance abuse; Homelessness; HIV risk behavior
MeSH Terms: conditions — Substance-Related Disorders | interventions — Case Management; Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CRA + HIV prevention (Experimental)
  Interventions: Behavioral: Community Reinforcement Approach (CRA) + HIV prevention
- Case Management + HIV prevention (Active Comparator)
  Interventions: Behavioral: Case Management + HIV Prevention
- MET + HIV prevention (Active Comparator)
  Interventions: Behavioral: Motivational Enhancement Therapy (MET) + HIV prevention

INTERVENTIONS:
Behavioral: Community Reinforcement Approach (CRA) + HIV prevention — 12 sessions of the CRA and 2 sessions of HIV prevention.
  Arms: CRA + HIV prevention
Behavioral: Case Management + HIV Prevention — 12 sessions of case management and 2 sessions of HIV prevention.
  Arms: Case Management + HIV prevention
Behavioral: Motivational Enhancement Therapy (MET) + HIV prevention — 2 sessions of MET and 2 sessions of HIV prevention.
  Arms: MET + HIV prevention

SUMMARY:
Youth who leave home for the streets are at significantly more risk for a multitude of problems, yet little research is available to guide treatment intervention efforts with this population. Studies document high rates of substance use, HIV risk, mental health problems, teenage pregnancy and criminality. Research to date examining homeless, street living youth has been primarily descriptive; less effort has been directed towards developing and evaluating treatment interventions for this group. The majority of homeless youth do not receive substance abuse treatment, with one study reporting that only 15% of street living youth report ever receiving mental health services. The effectiveness of the Community Reinforcement Approach (CRA) with street living youth was studied in our recently completed Stage 1 trial. The proposed study is a Stage II clinical trial examining outcome of CRA individual therapy as compared to two interventions commonly employed, yet little researched, with this group. All clients will be randomized to one of three theoretically distinct interventions: (1) CRA therapy, (2) Motivational Enhancement Therapy (MET), or (3) Case Management (CM). The relative effectiveness of these interventions will be evaluated at 3, 6, and 12 months post-baseline. The Social Ecology Theory of Development (Bronfenbrenner, 1979) guides our change hypotheses and intervention. Proposed change mechanisms (mediators) for each intervention will be evaluated. Differential treatment response as a function of ethnicity, gender, age, sexual orientation and abuse (moderators) will be investigated to better understand the interventions. The study will also examine how, if at all, treatment engagement, retention and expectations impact youth response to the three treatments. Information gained through this project may help address the gap in our understanding of how best to effectively intervene with a group at high risk for continuing health and psychological problems.

ELIGIBILITY:
Inclusion Criteria:

1. Youth are between the ages of 14-20.
2. Youth have plans to remain in the Columbus areas for at least 12 months.
3. Youth meets abuse or dependence DSM-IV criteria for Psychoactive Substance Use or Alcohol disorder, as assessed by the computerized diagnostic interview schedule for children (CDISC, Shaffer, 1992).
4. Youth agrees to participate in the assessment and treatment intervention.
5. Youth meets criteria for homelessness as defined by DHHS.

Exclusion Criteria:

1. Evidence of unremitted psychosis or other condition which would impair their ability to understand and participate in the intervention or consent for research participation (as determined by CDISC).

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 270 (Actual)
Dates: Start 2006-09; Primary Completion 2010-12 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Slesnick, Ph.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment ended on time, recruitment completed as proposed.
Pre-assignment Details: intent to treat design used.
Groups:
- CRA + HIV Prevention: Description of CRA: Treatment included twelve 1-hour sessions in addition to two HIV prevention sessions.
- MET + HIV Prevention: Description of MET: Treatment included two 1-hour sessions in addition to two HIV prevention sessions.
- Case Management + HIV Prevention: Description of CM: Treatment included twelve 1-hour sessions in addition to two HIV prevention sessions.
Period: Overall Study
Arm/Group | CRA + HIV Prevention | MET + HIV Prevention | Case Management + HIV Prevention
Started | 93 | 86 | 91
Completed | 93 | 86 | 91
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The number of participants in each group varies because the urn randomization program didn't balance the groups equally.
Groups:
- CRA + HIV Prevention; Case Management + HIV Prevention: Treatment included twelve 1-hour sessions for a total of 14 sessions.
- MET + HIV Prevention: Treatment included two 1-hour MI sessions for a total of 4 sessions
- Total: Total of all reporting groups
Arm/Group | CRA + HIV Prevention | MET + HIV Prevention | Case Management + HIV Prevention | Total
Number analyzed (Participants) | 93 | 86 | 91 | 270
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 16 | 10 | 43
  Between 18 and 65 years | 76 | 70 | 81 | 227
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 18.70 (1.34) | 18.69 (1.32) | 18.84 (1.11) | 18.7 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 37 | 47 | 127
  Male | 50 | 49 | 44 | 143
Region of Enrollment [Number; unit: participants]
  United States | 93 | 86 | 91 | 270

OUTCOME MEASURES:

1. Primary Outcome: Substance Use
Description: Percentage of substance use days in prior three months.
Time Frame: Three months
Population: The number of participants does not correspond to the participant flow model because some participants did not complete all follow-up assessment interviews. All available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: percent days of drug use
Groups:
- MET + HIV Prevention; Case Management + HIV Prevention: The number of participants does not correspond to the participant flow model because some participants did not complete all follow-up assessment interviews.
- CRA + HIV Prevention: The number of participants does not correspond to the participant flow model because some participants did not complete all follow-up assessment interviews. the groups equally.
Arm/Group | MET + HIV Prevention | CRA + HIV Prevention | Case Management + HIV Prevention
Number analyzed (Participants) | 66 | 70 | 66
percent days of drug use | 45.67 (43.24) | 53.60 (40.76) | 49.38 (40.66)

2. Secondary Outcome: HIV Risk
Description: Frequency of condoms use in prior three months.
Time Frame: Three months
Population: as for outcome 1
Measure: Number; unit: participants who always used condom
Groups:
- Case Management + HIV Prevention; CRA + HIV Prevention; MET + HIV Prevention: The number of participants does not correspond to the participant flow model because some participants did not complete all follow-up assessment interviews. All available data were included in the analysis.
Arm/Group | Case Management + HIV Prevention | CRA + HIV Prevention | MET + HIV Prevention
Number analyzed (Participants) | 58 | 66 | 57
participants who always used condom | 19 | 26 | 25

3. Secondary Outcome: HIV Risk
Description: Frequency of condoms use in prior three months.
Time Frame: Six months
Population: as for outcome 1
Measure: Number; unit: participants who always used condoms
Arm/Group | Case Management + HIV Prevention | MET + HIV Prevention | CRA + HIV Prevention
Number analyzed (Participants) | 58 | 62 | 65
participants who always used condoms | 25 | 29 | 25

4. Secondary Outcome: HIV Risk
Description: Frequency of condoms use in prior six months.
Time Frame: Twelve months
Population: as for outcome 1
Measure: Number; unit: participants who always used condoms
Arm/Group | Case Management + HIV Prevention | MET + HIV Prevention | CRA + HIV Prevention
Number analyzed (Participants) | 53 | 59 | 63
participants who always used condoms | 17 | 18 | 24

5. Secondary Outcome: Depressive Symptoms
Description: Beck Depression Inventory - II (BDI-II) total score, range from 0 (no depresion)to 63 (severe depression)
Time Frame: Three months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Case Management + HIV Prevention | CRA + HIV Prevention | MET + HIV Prevention
Number analyzed (Participants) | 66 | 70 | 66
units on a scale | 9.63 (9.57) | 14.78 (14.83) | 10.97 (12.20)

6. Secondary Outcome: Depressive Symptoms
Description: Beck Depression Inventory - II (BDI - II) Range from 0 (no depression) to 63 (severe depression)
Time Frame: Six months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Case Management + HIV Prevention | CRA + HIV Prevention | MET + HIV Prevention
Number analyzed (Participants) | 66 | 70 | 68
units on a scale | 10.02 (9.94) | 11.97 (14.13) | 8.76 (10.09)

7. Secondary Outcome: Depressive Symptoms
Description: Beck Depression Inventory - II (BDI-II) total score, range from 0 (no depression)to 63 (severe depression)
Time Frame: Twelve months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Case Management + HIV Prevention | CRA + HIV Prevention | MET + HIV Prevention
Number analyzed (Participants) | 64 | 71 | 69
units on a scale | 8.70 (11.09) | 12.07 (12.13) | 8.48 (10.93)

8. Primary Outcome: Substance Use
Description: Percentage of substance use days in prior three months
Time Frame: Six months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent days of drug use
Groups:
- CRA + HIV Prevention; MET + HIV Prevention; Case Management + HIV Prevention: The number of participants does not correspond to the participant flow model because some participants did not complete all follow-up assessment interviews. All available data were included int he analysis.
Arm/Group | CRA + HIV Prevention | MET + HIV Prevention | Case Management + HIV Prevention
Number analyzed (Participants) | 70 | 68 | 66
percent days of drug use | 39.10 (38.83) | 48.88 (41.43) | 42.64 (40.74)

9. Primary Outcome: Substance Use
Description: Percentage of substance use days in prior six months
Time Frame: Twelve months
Population: The number of participants does not correspond to the participant flow model because some participants did not complete all follow-up assessment interviews. All available data were included int he analysis.
Measure: Mean (Standard Deviation); unit: percent days of drug use
Arm/Group | MET + HIV Prevention | Case Management + HIV Prevention | CRA + HIV Prevention
Number analyzed (Participants) | 69 | 64 | 71
percent days of drug use | 49.25 (41.55) | 44.33 (39.31) | 38.46 (39.84)

ADVERSE EVENTS:
Time Frame: Overall Study
Description: Adverse events were monitored but none were observed.
Arm/Group | CRA + HIV Prevention | MET + HIV Prevention | Case Management + HIV Prevention
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/86 | 0/91
Other Adverse Events (participants affected / at risk) | 0/93 | 0/86 | 0/91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No